CLINICAL TRIAL: NCT04875767
Title: Cartilage Repair Using a Hyaluronic Acid-Based Scaffold With Bone Marrow Aspirate Compared With Microfracture for Focal Articular Cartilage Damage of the Hip: A Randomized Controlled Trial
Brief Title: Cartilage Repair Using a Hyaluronic Acid-Based Scaffold With Bone Marrow Aspirate Compared With Microfracture for Focal Articular Cartilage Damage of the Hip
Acronym: CHASE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding restrictions
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHASE01
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Femoroacetabular Impingement; Cartilage Damage
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors and those performing data entry and analysis will be blinded to the treatment allocation. Although patients will not be told which treatment they received, blinding may not be feasible given the intervention group will have an additional bone marrow harvest site incision at the iliac crest.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA-based scaffold with BMA (Hyalofast®; Anika Therapeutics, Bedford, MA, USA) (Experimental): Those allocated to the scaffold treatment group will have 30 ml of BMA harvested from the ipsilateral iliac crest under fluoroscopic guidance. The hip arthroscopy will then be resumed, and the damaged cartilage lesion will be debrided using a mechanical shaver to remove loose and calcified tissue. Once the walls of the lesion are confirmed to be stable with a probe, the exact size of the defect will be measured for templating of the scaffold. The biodegradable HA-based scaffold (Hyalofast®; Anika Therapeutics, Bedford, MA, USA) will be prepared by cutting it to fit the focal defect. Once the cartilage lesion is dried manually, this scaffold will be implanted into the defect after it has been soaked in the BMA. The scaffold will then be secured to the defect in a press-fit fashion to the surrounding cartilage. In the case where additional fixation of the scaffold is needed, such as uncontained shoulder of cartilage, fibrin glue will be used to secure the scaffold.
  Interventions: Device: HA-based scaffold with BMA (Hyalofast®; Anika Therapeutics, Bedford, MA, USA)
- Microfracture (Active Comparator): As per current standard of care for focal articular cartilage lesions of the acetabulum, the unstable cartilage will be debrided and removed from the subchondral bone using a mechanical shaver until a stable margin is obtained. A ring curette will be used to remove the calcified cartilage layer and create a border of healthy cartilage tissue that can support the marrow clot. Through the mid-anterior portal, specialized 90˚ awls will then be placed with the tip perpendicular to the subchondral bone of the acetabulum, and a mallet will be used to penetrate the subchondral bone with perforations 3 mm deep to access the bone marrow elements. This is done until the defect is homogeneously covered with micro-perforations 2-3 mm apart.
  Interventions: Device: HA-based scaffold with BMA (Hyalofast®; Anika Therapeutics, Bedford, MA, USA)

INTERVENTIONS:
Device: HA-based scaffold with BMA (Hyalofast®; Anika Therapeutics, Bedford, MA, USA) — General surgical and anaesthetic risks apply to the subjects included in the trial. Microfracture and BMA are surgical techniques currently being used and are approved for use in Canada. The HA-scaffold that will be used in this trial (Hyalofast®, Anika Therapeutics Inc.) has European CE Mark for use in all joints. We will obtain a Health Canada approval to use the Hyalofast® product in the hip for this trial.

SUMMARY:
Femoroacetabular impingement (FAI) is a hip disorder resulting from a mismatch of the hip joint, resulting in hip pain and can potentially cause osteoarthritis. As the head of the femur (ball of the hip) and the acetabulum (socket of the hip) impinge or rub together with this mismatch, patients can suffer damage to their articular cartilage which covers both. Currently, the standard of care to surgically treat articular cartilage damage is a procedure called 'microfracture' - where the surgeon makes multiple holes in the bone under the defects causing bone marrow cells and blood from the holes to combine to form a "super clot" that covers the damaged area and is meant to be the basis for new tissue formation or 'fibrocartilage'. However, native articular cartilage is made of hyaline, rather than fibrocartilage, which is a more flexible and durable tissue able to withstand a great deal of force on the hip when it moves. Therefore, a more recently developed strategy that has gained popularity for use in the repair of articular cartilage in the knee involves the implantation of bone marrow aspirate (BMA) along with a scaffold made of hyaluronic acid (HA) in a single-step procedure, with the goal of promoting new hyaline-like tissue. While this has shown promising results in treating knee cartilage damage, this treatment method has yet to be studied in the hip. This randomized controlled trial will evaluate in patients with painful articular cartilage damage of the hip, the effect of implantation of an HA scaffold along with BMA in comparison to microfracture on hip pain and function, cartilage regeneration, and any complications at 24 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-40 years
2. Hip pain lasting 6 months or more with no relief from documented non-operative modalities
3. Cam, Pincer, or Mixed FAI
4. Focal articular cartilage defects of the acetabulum on MRI, confirmed to be full thickness (International Cartilage Regeneration and Joint Preservation Society (ICRS) grade 3 or 4) during arthroscopic examination
5. Focal acetabular articular cartilage lesions measuring between 1x1 cm2 and 5x5 cm2 on MRI and confirmed on arthroscopic examination
6. Patient agrees to participate in the study-specific postoperative rehabilitation protocol
7. Patient can speak, read, and understand the language of the site
8. Patient has provided informed consent

Exclusion Criteria:

1. Cartilage defects of the femoral head
2. Previous surgery on the study hip
3. Traumatic chondral injury of the hip from a single event
4. Presence of advanced osteoarthritis (Tonnis grade 2 or 3)
5. Known hypersensitivity or allergy to hyaluronate
6. Evidence of hip dysplasia (i.e. lateral centre edge angle < 20˚)
7. Evidence of acetabular over coverage such as coxa profunda or coxa protrusion
8. Immunosuppressive or anti-proliferative medication use
9. Chronic pain syndromes
10. Significant medical co-morbidities (requiring assistance for activities of daily living (ADLs))
11. History of paediatric hip disease
12. Uncontrolled diabetes
13. Contraindications to MRI imaging (e.g. claustrophobia)
14. Patient is involved in ongoing legal or workplace claims
15. Patient is incarcerated
16. Patient who will likely have problems, in the judgement of the investigator, with maintaining follow-up

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
International Hip Outcome Tool-33 (iHOT-33) | 24 months
  The iHOT-33 is designed to measure hip-specific health-related quality of life changes after treatment of active young patients with hip disorders. The questionnaire has been validated in this patient population and has demonstrated efficacy, reliability, and responsiveness to change.

SECONDARY OUTCOMES:
Visual Analogue Scale (100-point scale) (VAS) | 24 months
  The VAS is one of the most frequently used pain rating scales in clinical practice and research. The VAS is a validated unidimensional scale that is easy to use, requires no verbal or reading skills, and is sufficiently versatile to be employed in a variety of settings.
Euro-Qol 5-D (EQ-5D) | 24 months
  The EQ-5D is a standardized, utility-based instrument for use as a measure of health outcome. It comprises 5 questions on mobility, self-care, usual activities, pain/discomfort, and anxiety/ depression. The EQ-5D has been used in previous studies involving patients with hip pain and has been extensively validated.
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | 24 months
  The MOCART scale has been validated to demonstrate the extent of cartilage restoration following surgical repair, examining factors such as "degree of defect repair and filling of the defect", and "integration to border zone". The MOCART scale is applied to MRIs.
Adverse events | 24 months
  Reported complications such as infection, additional or revision surgery, hypersensitivity or allergic reactions, reduced range of motion, and any other adverse events.

IPD SHARING:
Plan to Share IPD: No